CLINICAL TRIAL: NCT01326936
Title: Fast Track SBIR Study Online PCP Training in Screening, Brief Intervention, Referral, and Treatment
Brief Title: Online Primary Care Physician (PCP) Training in Screening, Brief Intervention, Referral, and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Directions, Inc (Industry)
Collaborators: University of Miami (Other); Cleveland Clinic Florida (Other); University of Arizona (Other); Contra Costa County Regional Medical Center (Unknown); Valley Family Medicine Residency, UC Davis Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R44DA026218 (NIH)
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Medical Education
Keywords: Online education; Medical education; Substance abuse training; Drug abuse training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unworked VP (Experimental): Online education using typical virtual patient (VP) approach. Five unworked VPs presented to subjects for study.
  Interventions: Behavioral: Online education
- Guided Learning (Experimental): Online education replaces two unworked VPs in Arm 1 with identical worked example VPs (case studies) for learners to study
  Interventions: Behavioral: Online education

INTERVENTIONS:
Behavioral: Online education — A brief (2-hour) interactive online training program in substance abuse (SU) management using virtual patient (VP) technology. Each learner will take one of two similar online programs involving five VPs that represent the range of SU management issues that commonly arise in clinical practice.

SUMMARY:
This project seeks to develop a comprehensive, computer-based education program for primary care physicians that will improve their skills in structured substance abuse screening, brief interventions, and referral and treatment (SBIRT). The investigators will develop two online education programs based on virtual patient (VP) technology. One program will include five typical, interactive, problem-solving VPs and the second will include five identical VPs except that two VPs will have been "worked" by substance abuse experts and presented as case studies. The remaining three VPs will be "unworked" (typical VPs). The investigators hypothesize that both education programs will significantly improve educational outcomes, compared to no training, as measured by a validated survey tool. A secondary hypothesis is that physicians using the "worked" (guided learning) program will achieve similar educational results as those using the typical VP approach, but will require less training time.

ELIGIBILITY:
Inclusion Criteria:

* Physician in primary care training program
* Faculty member in primary care training program

Exclusion Criteria:

* Advanced medical training in substance abuse management

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Scores on The Physicians' Competence in Substance Abuse Test (P-CSAT) | Following completion of education program and 2 months later
  The Physicians' Competence in Substance Abuse Test (P-CSAT) was developed as part of this project. Information, including a complete description of the P-CSAT, has been submitted for publication in a peer-reviewed journal

CONTACTS AND LOCATIONS:
Overall Officials: John M Harris, Jr., MD, Principal Investigator — Medical Directions, Inc
Locations (1):
- Medical Directions, Inc., Tucson, Arizona, United States

REFERENCES:
- [Result] Harris JM Jr, Sun H. The Physicians' Competence in Substance Abuse Test (P-CSAT): a multidimensional educational measurement tool for substance abuse training programs. Drug Alcohol Depend. 2012 May 1;122(3):236-40. doi: 10.1016/j.drugalcdep.2011.10.006. Epub 2011 Nov 4. PMID 22055011